CLINICAL TRIAL: NCT04599322
Title: Stabilometry Changes After Dry Needling in Flexor Digitoum Brevis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2706201911419 B
Record Dates: First submitted 2020-10-03; First posted 2020-10-22 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Healthy; Foot; Dry Needling
Keywords: Stabilometry; Dry needling; Trigger point

STUDY DESIGN:
Intervention Model Description: Pretest posttest of bilateral Flexor digitorum Brevis dry needling intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral dry needling in Flexor Brevis Digitorum in subjects with latent trigger point (Experimental): Bilateral dry needling in Flexor Brevis Digitorum in subjects with latent trigger point
  Interventions: Other: Bilateral dry needling in latent trigger points of the Flexor digitorum Brevis Muscle

INTERVENTIONS:
Other: Bilateral dry needling in latent trigger points of the Flexor digitorum Brevis Muscle — Bilateral dry needling in latent trigger points of the Flexor digitorum Brevis Muscle

SUMMARY:
The aim of this clinical trial is to check the balance effects of dry needling in the Flexor digitorum Brevis

DETAILED DESCRIPTION:
Eighteen healthy subjects wil be recruited for a quasi-experimental study. Participants will be from 18 to 40 years old, not obese. Participants will be measured before and after bilateral dry neddling in Flexor digitorum Brevis. The investigators will measure stabilometry variables with eyes open and closed.

Measures. Stabilometry will be measured by displacement of the center of pressures in X and Y with eyes open and closed , center of pressure (COP) with eyes open and closed, COP area with eyes open and closed, COP antero-posterior (a-p) and medio-lateral (m-lat) directions with eyes open and closed, and COP speed. Two trials will be recorded for each condition and the order of the conditions will be randomized across subjects, eyes open and eyes closed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Must have latent trigger point in Flexor Brevis Digitorum muscles

Exclusion Criteria:

* Previous lower extremities surgery.
* History of lower extremities injury with residual symptoms (pain, "giving-away" sensations) within the last year.
* Leg-length discrepancy more than 1 cm
* Balance deficits (determined by oral questionnaire regarding falls)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Stabilometry variable x displacement open eyes before dry needling | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with open eyes.
Stabilometry variable y displacement open eyes before dry needling | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with open eyes.
Stabilometry variable center of pressure area open eyes before dry needling | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes open.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction open eyes before dry needling | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction open eyes before dry needling | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).
Stabilometry variable x displacement before dry needling with closed eyes | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with eyes closed.
Stabilometry variable y displacement before dry needling with closed eyes | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with closed eyes.
Stabilometry variable center of pressure area before dry needling with closed eyes | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes closed.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction before dry needling with closed eyes | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction before dry needling with closed eyes | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).

SECONDARY OUTCOMES:
Stabilometry variable x displacement open eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with open eyes.
Stabilometry variable y displacement open eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with open eyes.
Stabilometry variable center of pressure area open eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes open.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction with open eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction with open eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).
Stabilometry variable x displacement with closed eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in milimeters) with eyes closed.
Stabilometry variable y displacement with closed eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in milimeters) with closed eyes.
Stabilometry variable center of pressure area with closed eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in milimeters²) with eyes closed.
Stabilometry variable center of pressure speed displacement of the anteroposterior(a-p) direction with closed eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in milimeters/second).
Stabilometry variable center of pressure speed displacement of the latero-lateral(lat-lat) direction with closed eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in milimeters/second).

CONTACTS AND LOCATIONS:
Overall Officials: Eva María Martínez-Jimenez, Principal Investigator — Mayuben Clinic
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvioli S, Guidi M, Marcotulli G. The effectiveness of conservative, non-pharmacological treatment, of plantar heel pain: A systematic review with meta-analysis. Foot (Edinb). 2017 Dec;33:57-67. doi: 10.1016/j.foot.2017.05.004. Epub 2017 Jun 15. PMID 29126045
- [Background] David JA, Sankarapandian V, Christopher PR, Chatterjee A, Macaden AS. Injected corticosteroids for treating plantar heel pain in adults. Cochrane Database Syst Rev. 2017 Jun 11;6(6):CD009348. doi: 10.1002/14651858.CD009348.pub2. PMID 28602048
- [Background] Salom-Moreno J, Sanchez-Mila Z, Ortega-Santiago R, Palacios-Cena M, Truyol-Dominguez S, Fernandez-de-las-Penas C. Changes in spasticity, widespread pressure pain sensitivity, and baropodometry after the application of dry needling in patients who have had a stroke: a randomized controlled trial. J Manipulative Physiol Ther. 2014 Oct;37(8):569-79. doi: 10.1016/j.jmpt.2014.06.003. Epub 2014 Sep 8. PMID 25199825
- [Background] Cotchett MP, Munteanu SE, Landorf KB. Effectiveness of trigger point dry needling for plantar heel pain: a randomized controlled trial. Phys Ther. 2014 Aug;94(8):1083-94. doi: 10.2522/ptj.20130255. Epub 2014 Apr 3. PMID 24700136
- [Background] McNally EG, Shetty S. Plantar fascia: imaging diagnosis and guided treatment. Semin Musculoskelet Radiol. 2010 Sep;14(3):334-43. doi: 10.1055/s-0030-1254522. Epub 2010 Jun 10. PMID 20539958